CLINICAL TRIAL: NCT05659641
Title: A Prospective, Multicenter, Open, Randomized Controlled, Non Inferiority Clinical Trial to Evaluate the Safety and Efficacy the Branch-based Intraoperative Stent System in the Treatment of Stanford A Aortic Dissection
Brief Title: The Branch-based Intraoperative Stent System in the Treatment of Stanford A Aortic Dissection（BROAD）
Acronym: BROAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Permed Biomedical Engineering Co., Ltd (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Fujian Medical University Union Hospital (Other); West China Hospital (Other); Changhai Hospital (Other); Yunnan Cardiovascular hospital (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); Anhui Provincial Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Southwest Hospital, China (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Linyi People's Hospital (Other); The First Hospital of Jilin University (Other); Second Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Hospital of Hebei Medical University (Other); The University of Hong Kong-Shenzhen Hospital (Other); Qilu Hospital of Shandong University (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS-CT（CN）
Record Dates: First submitted 2022-11-25; First posted 2022-12-21 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Aortic Dissection; Aneurysm, Dissecting; Aneurysm; Vascular Diseases; Cardiovascular Diseases
Keywords: Stanford A aortic dissection
MeSH Terms: conditions — Aortic Dissection; Aneurysm; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Learning Curve+Parallel+Single Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Branched Surgical Stent Graft System, (Experimental): Learning curve case group
  Experimental: Beijing PerMed Branched Surgical Stent Graft System,Permedos apex.
  Interventions: Device: PerMed Stent Graft System In Surgical Operation
- Single Branch Structure Stent Graft System single group (Experimental): Beijing PerMed single branch intraoperative stent system
  Interventions: Device: PerMed Stent Graft System In Surgical Operation
- CRONUS® Stent Graft System In Surgical Operation (Other): Control group：CRONUS® Stent Graft
  Interventions: Device: Endovastec CRONUS® Intraoperative stent system

INTERVENTIONS:
Device: PerMed Stent Graft System In Surgical Operation — PerMed Branch Stent Graft
  Other Names: Stanford A aortic dissection open surgery
  Arms: Branched Surgical Stent Graft System,; Single Branch Structure Stent Graft System single group
Device: Endovastec CRONUS® Intraoperative stent system — CRONUS® Branch Stent Graft
  Other Names: Stanford A aortic dissection open surgery
  Arms: CRONUS® Stent Graft System In Surgical Operation

SUMMARY:
The purpose of the study was to evaluate the safety and efficacy of a branched type intraoperative stent system for the treatment of Stanford type A aortic dissection

DETAILED DESCRIPTION:
Types The clinical trial design was prospective, muticenter, open, randomized controlled design with an additional single group design.

Plan Before the randomized controlled trial, each center will enroll one subject as a learning curve case（only use PerMed double branched structures）. 212 participants were planned to be enrolled from no less than 10 qualified clinical research institutions and randomly assigned 1:1 to the intraoperative stent systems of Endovastec and the branched type intraoperative stent systems of PerMed double branched structures. An additional 30 subjects were enrolled using a branched type intraoperative stent system with a single branch structure from PerMed, Beijing.

All enrolled participants were followed up clinically intraoperatively, before discharge or 30 days ± 7 days after procedure, 6 months ± 30 days after procedure, 12 months ± 30 days after procedure, and 2-5 years after procedure.Non inferiority of the trial product to the control product was assessed with the primary end point of all-cause mortality at 12 months after procedure. The statistical analysis and summary report will be conducted based on the 12-month follow-up data of all subjects, and the application for medical device registration will be carried out. The long-term efficacy and safety evaluation of the product will be carried out after long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years, male or female;
2. Stanford type A aortic dissection subjects with involvement of the descending arch aorta；
3. Subjects treated with stent pictorial procedures as judged appropriate by the investigator；
4. Subjects or their legal surrogates were able to understand the purpose of the study, had adequate compliance to the clinical study protocol, and voluntarily signed the informed consent form.

Exclusion Criteria:

1. Subjects with aortic dissections confined to the ascending and / or arch
2. Subjects with a left common carotid artery branch vessel diameter < 5 mm or > 16 mm (not applicable to subjects enrolled with a single branch structure)
3. Subjects with a left subclavian artery branch vessel diameter < 7 mm or > 16 mm
4. Subjects with aortic dissection with severe malperfusion syndrome preoperatively (e.g., subjects presenting with coma, paraplegia, need for dialysis, gastrointestinal necrosis or limb necrosis due to ischemia, etc.)
5. Subjects with vertebral artery variants
6. Subjects with infectious aortic dissections
7. Subjects with acute systemic infection, severe infection and associated sepsis, shock or multiple organ failure
8. Subjects unable to tolerate anaesthesia and cardiopulmonary bypass
9. Subjects who had undergone open surgical procedures of the cardiocerebral vasculature within 90 days prior to surgery
10. Subjects with history of active bleeding, coagulopathy or refusal of blood transfusion
11. Subjects known to be allergic to materials such as contrast agents, nitinol alloys, coated artificial blood vessels
12. Subjects with a life expectancy of less than 12 months (other than disease due to aortic dissection)
13. Subjects being enrolled in other clinical trials
14. Pregnant and lactating women, and subjects with a recent pregnancy preparation
15. Subjects with poor compliance other conditions that the investigator considers inappropriate for participation in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | after procedure 1 year
  Percentage of subjects who died from any cause within 12 months ±30 days

SECONDARY OUTCOMES:
Device implantation success rate | Immediately after implantation
  Refers to the proportion of successful device implantation. That is, the test product or control product was successfully introduced into the true lumen of the vessel and successfully released, the delivery system was successfully withdrawn, and the anastomosis was completed with the artificial vessel.
Operation success rate | Immediately after procedure
  It refers to the proportion of subjects who have completed the expected surgical treatment
30 day all-cause mortality after procedure | 30 day
  It refers to the proportion of dead subjects within 30 days (including 30 days) after operation
false-lumen thrombosis rates | 6 month, 1 year
  Complete thrombosis refers to the rate of complete thrombosis of the entire aortic false lumen on arterial phase and delayed phase imaging.
  Partial thrombogenicity refers to the rate of presence of thrombus in the false lumen but residual flow in the arterial and delayed phases. Details are described in the 2022 ACC guidelines for the diagnosis and management of AHA aortic disease.
Branch patency | 1 year
  The proportion of subjects with stenosis degree of left subclavian artery and/or left common carotid artery less than 50% within 12 months after procedure.
Secondary intervention rate of target lesions | 1 year
  The proportion of participants with unexpected re intervention due to the trial or control device.
stroke rate | 1 year
  It refers to a cerebrovascular event caused by the implantation of the test product or control product, which shows partial or complete loss of movement or sensation, and lasts for more than 24 hours
Incidence of spinal cord ischemia | 1 year
  It refers to the ratio of subjects with spinal cord functional defects caused by ischemia after the implantation of the experimental or control device. Except those caused by tumor, trauma, tuberculosis and other factors with clear causes
Incidence of acute kidney injury | 1 year
  Renal hypofunction refers to the increase of serum creatinine (SCR) ≥ 50% compared with the basic value (SCR value in screening period) and (or) urine volume<0.5 ml/(kg · h)>6 h. Except for acute renal injury caused by poisoning and other clear causes.
Mortality associated with aortic dissection | 30 day
  It refers to the proportion of subjects who died of aortic dissection within 30 days (inclusive) after operation or within 30 days (inclusive) after the secondary intervention of target lesion
Incidence of device-related adverse events | 6month，1 year，5 year
  It refers to the ratio of device related adverse events occurring after the implantation of the test product in the follow-up period to the total adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Chunsheng Wang, Dr, Principal Investigator — Shanghai Zhongshan Hospital
Locations (18):
- China (18):
  - Anhui Provincial Hospital, Hefei, Anhui
  - First Hospital Affiliated to the Army Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Wuhan Union Hospital, China, Wuhan, Hubei
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital Xi'an Jiaotong University, Xi'an, Shaanxi
  - Linyi People's Hospital, Linyi, Shandong
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Shenzhen
  - West China Hospital, Chengdu, Sichuan
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yan 'an Hospital Affiliated to Kunming Medical University, Kunming, Yunnan
  - Permed Biomedical Engineering Co., Ltd, Beijing

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT05659641/ICF_000.pdf